CLINICAL TRIAL: NCT01280409
Title: The Effects of Metformin on Retained Postpartum Weight in Women With Gestational Diabetes: A Randomized, Placebo-Controlled Trial
Brief Title: Metformin Postpartum for GDM RCT for Reduced Weight Retention
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Gilstrap, Larry C, M.D. (Individual)
Responsible Party: Principal Investigator, Jerrie Refuerzo, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC-MS-10-0426
Record Dates: First submitted 2011-01-19; First posted 2011-01-20 (Estimated); Results first posted 2018-11-28 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Diabetes, Gestational
MeSH Terms: conditions — Diabetes, Gestational | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Compounded placebo
  Interventions: Drug: Placebo
- Metformin (Experimental): Compounded metformin as the intervention
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Subjects will receive metformin 850 mg PO daily for 7 days, then metformin 850mg PO twice a day for the next 5 weeks
  Arms: Metformin
Drug: Placebo — Subjects will receive a placebo (similar in size, taste, color) once daily for 7 days, then twice daily for the next 5 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether the study drug metformin is helpful in reducing weight after pregnancy in women with gestational diabetes. This pilot study will provide information on how well women are able to take metformin postpartum, whether metformin increases weight loss, and whether there are any increased risks of side effects to you as a new mother.

DETAILED DESCRIPTION:
At 24-48 hours after delivery, women who are eligible for participation will be approached and consented to the study. Maternal weight will be measured and 20ml of maternal blood will be obtained to assess glucose control and lipid profile. Women will be counseled regarding diet, exercise and glucose control. Data including maternal demographics, clinical characteristics and neonatal outcomes will be collected. At 3 weeks postpartum, a research nurse will contact the subject via telephone call to inquire about adverse or side effects, ability to take the prescribed medication (metformin or placebo), and to answer questions about the study. At 6 weeks postpartum, maternal weight will be measured , blood will be obtained and side effects will be evaluated again. Finally, a satisfaction survey will be completed.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum women with a delivery greater than 34 weeks of pregnancy
* Between the ages of 18 to 49 years
* Women with a diagnosis of gestational diabetes mellitus (either treated with insulin, oral hypoglycemic agent or diet-controlled) after 24 weeks in most recent pregnancy based on a confirmatory 3 hour glucola test (based on either the Carpenter and Coustan's of the Diabetes Task Force criteria)

Exclusion Criteria:

* women with pre-gestational diabetes mellitus (either Type I or Type II DM)
* women unable to tolerate metformin based on patient history
* women who will be discharged hom eon insulin or oral hypoglycemic agent in the immediate postpartum period
* women with a BMI <25 kg/m²

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2011-01; Primary Completion 2014-03 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerrie S Refuerzo, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (2):
- United States (2):
  - Memorial Hermann Hospital, Texas Medical Center, Houston, Texas
  - University of Texas Health Science Center at Houston, Professional Building, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Metformin
Started | 59 | 55
Completed | 43 | 36
Not Completed | 16 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Metformin | Total
Number analyzed (Participants) | 43 | 36 | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 43 | 36 | 79
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.8 (6.4) | 31.6 (5.3) | 30.2 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 36 | 79
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 43 | 36 | 79

OUTCOME MEASURES:

1. Primary Outcome: Weight Change
Description: The weight change in kilograms defined as:
  weight change = Weight(pp) - Weight(6wk)
Time Frame: within 24 hours after delivery; at 6 weeks postpartum visit (2nd research visit)
Measure: Median (Full Range); unit: kg
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 43 | 36
kg | 6.5 [-0.3 to 12.1] | 6.3 [-0.3 to 19.8]

2. Secondary Outcome: Number of Participants Who Achieved Pre-pregnancy Weight
Time Frame: At 6 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 43 | 36
Participants | 16 | 15

3. Secondary Outcome: Number of Participants Who Achieved Their Ideal Body Weight
Time Frame: At 6 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 43 | 36
Participants | 1 | 1

4. Secondary Outcome: Hemoglobin a1c
Description: We will calculate the change in hemoglobin a1c.
Time Frame: At 6 weeks postpartum
Population: This data is not reported because blood samples were not analyzed for Hemoglobin a1c.
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: HDL, LDL, Triglyceride
Description: We will calculate the change in LDL, HDL, and triglyceride levels.
Time Frame: At 6 weeks postpartum
Population: This data is not reported because blood samples were not analyzed for HDL, LDL, and triglyceride.
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Self-reported Compliance With Medications
Time Frame: 3 weeks postpartum
Population: 46 in the placebo group and 53 in the metformin group were available by phone at 3 weeks postpartum to indicate medication compliance.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 46 | 53
Participants
  Unknown | 1 | 4
  less than 50% | 12 | 10
  greater than 50% | 19 | 20
  100% | 14 | 19

7. Secondary Outcome: Self-reported Compliance With Medications
Time Frame: 6 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 43 | 36
Participants
  Unknown | 0 | 0
  less than 50% | 1 | 1
  greater than 50% | 14 | 18
  100% | 28 | 17

8. Secondary Outcome: Difficulty With Diet as Assessed by a 5-point Likert Scale
Time Frame: At 6 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 43 | 36
Participants
  Not at all | 10 | 9
  Slightly | 9 | 10
  Moderately | 14 | 14
  Quite | 6 | 1
  Extremely | 4 | 2

9. Secondary Outcome: Difficulty With Exercise as Assessed by a 5-point Likert Scale
Time Frame: At 6 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 43 | 36
Participants
  Not at all | 11 | 11
  Slightly | 9 | 6
  Moderately | 13 | 13
  Quite | 4 | 5
  Extremely | 6 | 1

10. Secondary Outcome: Difficulty With Medication as Assessed by a 5-point Likert Scale
Time Frame: At 6 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 43 | 36
Participants
  Not at all | 15 | 14
  Slightly | 7 | 6
  Moderately | 5 | 7
  Quite | 6 | 5
  Extremely | 10 | 4

11. Secondary Outcome: Satisfaction With Diet as Assessed by a 5-point Likert Scale
Time Frame: At 6 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 43 | 36
Participants
  Not at all | 2 | 6
  Slightly | 5 | 7
  Moderately | 9 | 8
  Quite | 12 | 11
  Extremely | 15 | 4

12. Secondary Outcome: Satisfaction With Exercise as Assessed by a 5-point Likert Scale
Time Frame: At 6 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 43 | 36
Participants
  Not at all | 3 | 6
  Slightly | 9 | 6
  Moderately | 14 | 14
  Quite | 9 | 6
  Extremely | 8 | 4

13. Secondary Outcome: Satisfaction With Medication as Assessed by a 5-point Likert Scale
Time Frame: At 6 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 43 | 36
Participants
  Not at all | 4 | 5
  Slightly | 6 | 4
  Moderately | 6 | 7
  Quite | 11 | 11
  Extremely | 16 | 9

ADVERSE EVENTS:
Time Frame: 3 weeks postpartum
Arm/Group | Placebo | Metformin
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/46
Other Adverse Events (participants affected / at risk) | 7/56 | 12/46
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=56) | Metformin (N=46)
Nausea (Gastrointestinal disorders) | 7 (7) | 7 (7)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 6 (6) | 8 (8)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (3) | 4 (4)
Medication Intolerance (General disorders) | 5 (5) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No